CLINICAL TRIAL: NCT06862856
Title: A Prospective Study of Flotufolastat F 18 Positron Emission Tomography in Men With Very Low Prostate Specific Antigen Recurrence
Brief Title: Flotufolastat F 18 PET in Men With Very Low PSA Recurrence
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Principal Investigator, Jason Efstathiou, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 24-770
Record Dates: First submitted 2025-02-20; First posted 2025-03-06 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer (Adenocarcinoma); Prostate Specific Antigen
Keywords: flotufolastat F 18 positron emission tomography; low prostate specific antigen recurrence; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Very Low Prostate Specific Antigen Recurrence: Men >18 years of age will undergo screening to confirm eligibility for this research study. Participants will receive a PET scan with flotufolastat F 18 injection on study visit 2.
  Interventions: Diagnostic Test: Positron Emission Tomography (PET)

INTERVENTIONS:
Diagnostic Test: Positron Emission Tomography (PET) — This is a PET scan with flotufolastat F 18 injection.
  Other Names: Flotufolastat F 18 PET

SUMMARY:
The purpose of this study is to assess detection rate of flotufolastat F 18 positron emission tomography (PET) for low prostate specific antigen (PSA) recurrence of prostate cancer (PC) following radical prostatectomy.

DETAILED DESCRIPTION:
This is a prospective single arm study for the use of flotufolastat F 18 PET in men with very low prostate specific antigen recurrence. The research study involves collecting flotufolastat F 18 PET images to evaluate the detection rate. Flotufolastat F 18 is a radiopharmaceutical (radioactive agent) the U.S. Food and Drug Administration (FDA) has approved. Participation in this study will be for the duration of the flotufolastat F 18 PET scan. It is expected that about 50 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a history of localized histologically confirmed adenocarcinoma of the prostate and have received radical prostatectomy (RP) with curative intent.
* Participants must have measurable disease, defined as a non-zero PSA value post-RP that is concerning for biochemically recurrent or persistent disease, is ≤0.20 ng/mL, and obtained within 60 days of PET/CT.
* At least 6 weeks must have elapsed after RP. If previously taking ADT, it should have been discontinued at least 16 weeks prior to PET.
* Participants with a clinical flotufolastat F 18 PSMA PET/CT scan prescribed as part of the standard of care management.
* Age ≥18 years.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants currently receiving ADT (defined as surgical orchidectomy; luteinizing hormone-releasing hormone [LHRH] agonist alone [continuous or intermittent]; LHRH antagonist alone [continuous or intermittent]; administration or use of a first or second generation anti-androgen alone or in combination with an LHRH agonist/antagonist).
* Participants who are receiving any other investigational agents for this condition within five biological half-lives prior to administration of flotufolastat F 18.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to flotufolastat F 18 or other agents used in study.
* Participants receiving any of the following substances will be considered ineligible: x-ray contrast agent <24 hours prior to the flotufolastat F 18 PET and any other PET imaging agent within 24 hours or 10 half-lives, whichever is longer, prior to the flotufolastat F 18 PET/CT. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men of all races and ethnic groups are eligible for this trial
Study Population: Participants will be identified and screened for eligibility via physician referral, clinic visit, or medical record review.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Detection Rate | Periprocedural to date of detected lesion
  The detection rate is defined as the percentage of all patients scanned who have at least one positive lesion (localized correspondence between flotufolastat F 18 PET/CT imaging and the reference standard) regardless of coexisting false positive findings.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Efstathiou, MD, DPhil, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Jason Efstathiou, MD, DPhil (efstathiou@mgb.org) at 617-726-5866. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation